CLINICAL TRIAL: NCT00401505
Title: Rubella Susceptibility in Multiparous Women
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 06-186
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Rubella; Vaccine
Keywords: rubella; rubella vaccine; postpartum; immunity
MeSH Terms: conditions — Rubella

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine the reasons why multiparous women (women who are pregnant and have been pregnant before) might still be susceptible to rubella.

DETAILED DESCRIPTION:
This study is designed to investigate why multiparous women might still be susceptible to rubella. All pregnant women are checked for rubella immunity, and if they are non-immune, there are standard orders in our hospital to administer the rubella vaccine on the post-partum floor prior to discharge home from the hospital. Despite this, some multiparous women are found to be susceptible (non-immune), and this study will explore the reasons for this.

ELIGIBILITY:
Inclusion Criteria:

* All rubella susceptible women who delivered during the study period.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All rubella susceptible women who delivered during the study period.
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2006-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Yudin, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada